CLINICAL TRIAL: NCT00699465
Title: A Double-blind Randomized Trial to Compare the Efficacy of Intermittent Pneumatic Compression (IPC) With and Without Early Anticoagulant Treatment for Prevention of Venous Thromboembolism (VTE) in Patients With Acute Primary Intracerebral Hemorrhage (ICH)
Brief Title: Prevention of Venous Thromboembolism in Patients With Acute Primary Intracerebral Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Oulu University Hospital (Matti Hillbom), Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EUDRACT 2007-006206-24
Record Dates: First submitted 2008-06-12; First posted 2008-06-18 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: Thromboprophylaxis; Prevention of venous thromboembolism after ICH; Enoxaparin; Intermittent pneumatic compression
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Early enoxaparin
  Interventions: Drug: enoxaparin
- 2 (Placebo Comparator): Late enoxaparin
  Interventions: Drug: enoxaparin placebo

INTERVENTIONS:
Drug: enoxaparin — 20 mg enoxaparin (2 000 IU) s.c. will be given twice daily starting 24-48 h after onset of the stroke. Intermittent pneumatic compression will be started immediately after admission.
  Other Names: Klexane; Kendall
  Arms: 1
Drug: enoxaparin placebo — Placebo will be given s.c. twice daily starting 24-48 h after onset of the stroke for 2 days. Thereafter, 20 mg enoxaparin (2 000 IU) s.c. will be given twice daily. Intermittent pneumatic compression will be started immediately after admission.
  Other Names: Klexane; Kendall
  Arms: 2

SUMMARY:
* To evaluate the efficacy of using IPC during the acute phase of ICH in the prevention of VTE.
* To assess the safety and efficacy of additional therapy with enoxaparin.
* To compare the efficacy and safety of the European and American guideline recommendations.
* To provide an efficient and safe thromboprophylaxis for several weeks until the patient is able to walk.

DETAILED DESCRIPTION:
* Although it has been poorly investigated, the risk of VTE among patients with acute primary intracerebral hemorrhage is generally believed to be at least as high as among patients with ischemic stroke.
* The currently available guidelines state that while low doses of subcutaneous heparin or low-molecular-weight heparin may reduce VTE, it is possible that their effect is counterbalanced by an increase in hemorrhagic complications.
* It is still unclear when (if ever) low-molecular-weight-heparin should be safely initiated in ICH patients.

ELIGIBILITY:
Inclusion Criteria:

* acute primary ICH
* > 17 years
* unable to walk
* admitted within 12 h after onset of ICH
* informed consent obtained

Exclusion Criteria:

* other type of ICH than acute primary intracerebral hemorrhage
* patients who need neurosurgery
* evidence of VTE at screening
* thrombolytic treatment within the preceding week
* major surgery or major trauma within the preceding 3 months
* life expectancy less than 3 months due to comorbid disorders
* confirmed malignant disease (cancer)
* hepatitis and/or liver cirrhosis
* renal failure
* infectious disease (HIV, endocarditis etc.)
* current of previous hematologic disease
* recent active and untreated gastric/duodenal ulcer
* allergy or known hypersensitivity to enoxaparin or heparins
* known hypersensitivity to benzyl alcohol
* women of childbearing age if pregnant
* participation in another study within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The cumulative occurrence of confirmed VTE, defined as the composite of symptomatic or asymptomatic DVT, or symptomatic or fatal PE occurring during the treatment period. | 90 days

SECONDARY OUTCOMES:
Bleeding complications including rebleedings occurring within the treatment period | 90 days
Increase in ICH volume observed by head CT or at autopsy during the treatment period | 90 days
Cardiovascular death occurring within the treatment period | 90 days
Death due to any cause occurring within the treatment period | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Matti E Hillbom, MD, PhD, Study Chair — Oulu University Central Hospital, Department of Neurology; Seppo S Juvela, MD, PhD, Study Director — Turku University Central Hospital, Department of Neurosurgery; Turgut Tatlisumak, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Department of Neurology; Liisa K Luostarinen, MD, PhD, Principal Investigator — Päijät-Häme Central Hospital, Department of Neurology; Aimo Rissanen, MD, PhD, Principal Investigator — Keski-Suomen Keskussairaala; Heikki Numminen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Department of Neurology, Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Background] Steiner T, Kaste M, Forsting M, Mendelow D, Kwiecinski H, Szikora I, Juvela S, Marchel A, Chapot R, Cognard C, Unterberg A, Hacke W. Recommendations for the management of intracranial haemorrhage - part I: spontaneous intracerebral haemorrhage. The European Stroke Initiative Writing Committee and the Writing Committee for the EUSI Executive Committee. Cerebrovasc Dis. 2006;22(4):294-316. doi: 10.1159/000094831. Epub 2006 Jul 28. PMID 16926557
- [Background] Broderick J, Connolly S, Feldmann E, Hanley D, Kase C, Krieger D, Mayberg M, Morgenstern L, Ogilvy CS, Vespa P, Zuccarello M; American Heart Association; American Stroke Association Stroke Council; High Blood Pressure Research Council; Quality of Care and Outcomes in Research Interdisciplinary Working Group. Guidelines for the management of spontaneous intracerebral hemorrhage in adults: 2007 update: a guideline from the American Heart Association/American Stroke Association Stroke Council, High Blood Pressure Research Council, and the Quality of Care and Outcomes in Research Interdisciplinary Working Group. Stroke. 2007 Jun;38(6):2001-23. doi: 10.1161/STROKEAHA.107.183689. Epub 2007 May 3. PMID 17478736